CLINICAL TRIAL: NCT04014712
Title: Role of Nitric Oxide Coupling in Muscle Dysfunction With COPD
Brief Title: O2 Transport and Utilization in Health and Lung Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit due to COVID-19 pandemic
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-4815
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: COPD; Tetrahydrobiopterin Deficiency; Oxidative Stress
Keywords: BH4; Exercise; Mitochondria; Vascular function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Phenylketonurias; Motor Activity | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- acute BH4/Tetrahydrobiopterin treatment (Experimental): Oral supplement, Pill, 10 mg/kg of body weight
  Interventions: Drug: Tetrahydrobiopterin
- Placebo (Placebo Comparator): Oral supplement, Pill, Placebo pill with inert excipient
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tetrahydrobiopterin — Oral, Single dose
  Arms: acute BH4/Tetrahydrobiopterin treatment
Drug: Placebo oral tablet — Single dose
  Arms: Placebo

SUMMARY:
Skeletal muscle dysfunction is a frequent and clinically relevant systemic manifestation of Chronic Pulmonary Obstructive Disease (COPD), which is still poorly understood. Therefore, the focus of this study is on the role of a deficit in tetrahydrobiopterin and nitric oxide synthase uncoupling induced by chronic oxidative stress on metabolic and vascular abnormalities in skeletal muscle of patients suffering from COPD.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of supplementation with tetrahydrobiopterin (BH4) for improving vascular and muscle function in patients with COPD and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be between the age of 18 and 85 years;
* For the COPD cohort, patients with a diagnosis of stable COPD (i.e., those not experiencing an acute exacerbation of symptoms) and spirometric evidence of airway obstruction (FEV1 <80% predicted, FEV/FVC<0.70);
* Ability to perform motor tests;
* Ability to provide informed consent

Exclusion Criteria:

* uncontrolled hypertension;
* hyperlipidemia;
* recent exacerbation;
* Major cardiovascular event procedure (<3 months);
* Pregnancy
* known significant hepatic, renal disease, active substance abuse
* contraindication to MRI, claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function | 4 hours
  PCr recovery kinetics
intracellular PO2 | 4 hours
  Myoglobin oxygenation

SECONDARY OUTCOMES:
systemic blood markers of oxidative stress | 4 hours
  blood markers
Peripheral Blood flow | 4 hours
  Exercise Blood flow by Doppler Ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Applied Life Sciences, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months post-publication
Access Criteria: Within 6 months after the data have been published, and upon written request, a limited, de-identified, anonymized dataset will be created pursuant to the Data use Agreement.